CLINICAL TRIAL: NCT05107466
Title: Quantification of Visually Evoked Cortical Potentials in Individuals With Hearing Loss
Status: Recruiting | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Dartmouth College (Other)
Responsible Party: Principal Investigator, James E. Saunders, Professor of Otology and Neurotology, Department of Otolaryngology, Dartmouth-Hitchcock Medical Center
Other Study IDs: STUDY02001061
Record Dates: First submitted 2021-10-25; First posted 2021-11-04 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Sensorineural Hearing Loss; Hearing Loss
Keywords: cochlear implant
MeSH Terms: conditions — Hearing Loss, Sensorineural; Hearing Loss

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Individuals with Hearing Loss: 60 adults (>18 y/o) with a diagnosis of hearing loss. These participants may use cochlear implant(s), hearing aid(s), or have unaided hearing loss.
  Interventions: Diagnostic Test: P300 Visually evoked potential
- Individuals with Normal Hearing: 40 adults (>18 y/o) without a diagnosis of hearing loss.
  Interventions: Diagnostic Test: P300 Visually evoked potential

INTERVENTIONS:
Diagnostic Test: P300 Visually evoked potential — Measurement of the late cortical response, P300 potential to visually evoked stimuli using an oddball paradigm.

SUMMARY:
This research is being done to determine whether a test that measures a "Visual Evoked Potential" can be used in a new way for individuals that have hearing loss. This test measures the participant's brain's response (so called "brain waves") to specific visual images. This study will help the investigators determine whether this test could be used to improve treatments for patients with hearing loss.

The "Visual Evoked Potential" measurement test is already used in the investigator's Neurology clinic at Dartmouth Hitchcock Medical Center for various conditions to measure "early" brain responses that occur in the first 1-2 seconds after a new cue. Our research aims to explore your brain's response just after that early 1-2 second period by looking at a specific response called the "P300". The P300 wave is a brain response to new or different images or sounds. A visual evoked P300 has not been studied in individuals with hearing loss.

The investigators will compare the results of this test to standard auditory tests, tests of cognitive function, and cochlear implant patient outcomes to explore how these factors can predict successful use of a hearing aid or cochlear implant.

DETAILED DESCRIPTION:
Participants will schedule two appointments, at times convenient to the participant, to come to the testing clinic to complete the Visual Evoked Potential testing as well as the auditory test, cognitive/mood assessment battery, and sound quality survey included in this study.

The first research appointment will include a test of the participant's vision that involves looking at a chart on a wall and identifying appropriate letters. After this brief visual test, the participant will complete VEP testing.

For the VEP portion of the testing, participants will sit in a comfortable chair and have electrodes placed at several locations on their scalp. Electrodes are stickers that connect to a wire that connects to a computer. Electrodes do not break the skin or commonly cause any discomfort or harm. Participants will sit for approximately 1 hour and watch images presented to them on a computer screen while the participant's brain's response is measured using a computer. A picture of the electrodes on the participant's head will be taken for precise electrode localization.

The second research appointment will consist of an auditory test, a cognitive/mood assessment, and a cochlear implant sound quality survey. The survey will only be completed by participants with a cochlear implant. The auditory testing portion will take place in the Audiology clinic and requires participants to listen and respond to different patterns of sound. While participants are at the clinic for testing, they will be asked to complete several questionnaires that ask about participant's mood and thought processing. Participants with cochlear implants will also be asked to complete a questionnaire about their perceived sound quality with their implant(s).

The Visual Evoked Potential measure, auditory test results, cognitive/mood assessment, and cochlear implant sound quality survey responses will be compared between "hearing loss" and "normal hearing" groups to determine if VEP testing can be used in a new way to predict successful use of a cochlear implant or hearing aid.

ELIGIBILITY:
Inclusion

* Subjects will be recruited from the Otolaryngology/Audiology clinic at DHMC with the goal of enrolling subjects with a variety of degrees of hearing loss and central auditory processing dysfunction.
* Age > 18 y/o.
* Current and new patients receiving care in the DHMC Otolaryngology clinic or from the employees of Dartmouth College, DHMC, and the community, will be included as allowed under COVID guidelines.

Exclusion

* Patients with known brain pathology (e.g., CNS tumors, CVA diagnosis, etc…) will be excluded.
* Patients with severe neurological or neuropsychological disorders will be excluded.
* Patients with known seizure history will be excluded.
* Patients with known blindness will be excluded.
* The following special populations will not be included:
* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults (>18 y/o) with or without a diagnosis of hearing loss.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-07-28 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Difference in mean VEP latency as measured by onset time of the P300 wave from time of stimuli presentation. | 30 minutes
  Difference in P300 VEP latency to odd ball paradigm visual stimuli in individuals with hearing loss and normal hearing controls. Differences in VEP latency will be measured by recording onset time of the P300 signal from time of stimuli presentation.
Difference in mean VEP amplitude as measured by the maximum voltage reached by the P300 wave after presentation of stimulus before returning back to zero. | 30 minutes
  Difference in mean VEP amplitude to odd ball paradigm visual stimuli in individuals with hearing loss and normal hearing controls. Differences in VEP amplitude will be measured by recording maximum voltage reached by the P300 wave after presentation of stimulus before returning back to zero.

SECONDARY OUTCOMES:
Difference in Gap Detection Thresholds as a measure of auditory processing. | 15 min
  Difference in Gap Detection Thresholds between individuals with hearing loss and normal hearing controls. Thresholds (in ms) will be measured and calculated using a software developed by a local engineering company (Creare) in a DHMC Audiology clinic sound booth.
Difference in cochlear implant sound quality perception as measured by survey responses from participants with cochlear implants. | 10 min
  Participants with cochlear implants will be asked to complete a subjective survey to provide detail about their experience with cochlear implant(s). The survey responses contain both multiple choice answers and continuous rating scales to allow participants to answer questions pertaining to their perception of music, voices, meditative sounds, and general sound perception. The survey is not a scored on a scale, but is instead meant to capture a participant's unique, subjective perception of sound.
Difference in scores for the Repeatable Battery for the Assessment of Neuropsychological Status for Hearing-impaired individuals (RBANS-H) between individuals with hearing loss and normal hearing controls. | 45 minutes
  The RBANS-H is a cognitive assessment battery that consists of the 12 following items: List Learning, Story Memory, Figure Copy, Line Orientation, Picture Naming, Semantic Fluency, Digit Span, Coding, List Recall, List Recognition, Story Recall, and Figure Recall. The minimum (worst) RBANS-H score is 0 and the maximum (best) RBANS-H score is 321.
Difference in completion times for the Trail Making Test between individuals with hearing loss and normal hearing controls. | 5 min
  The Trail Making Test is a standard neuropsychological assessment that requires a pen and paper. Part A requires that participants connect randomly placed numbers in ascending order. Part B requires that participants connect randomly placed numbers and letters in alternating numerical/alphabetical order. The Trail Making Test is scored by time (i.e. minutes:seconds). Faster completions of the test are better outcomes than slower completions.
Difference in Controlled Oral Word Fluency Test scores between individuals with hearing loss and normal hearing controls. | 5 min
  The Controlled Oral Word Fluency Test is a standard neurocognitive assessment. Participants are given one minute to generate as many words as possible that start with a given letter of the alphabet. Better scores reflect a higher number of words provided, and worse scores reflect fewer words provided by the participant.
Difference in scores for the Test of Premorbid Functioning between individuals with hearing loss and normal hearing controls. | 5 min
  The Test of Premorbid Functioning is a standard neurocognitive assessment that requires participants to read aloud from a list of pre-selected words. The total score is the number of words that the participant pronounces correctly. The minimum (worst) score for this assessment is 0, and the maximum (best) score is 70.
Difference in scores for the Beck Depression Inventory-II (BDI-II) between individuals with hearing loss and normal hearing controls. | 5 min
  The Beck Depression Inventory-II is a standard depression scale. This assessment is a survey that contains 21 multiple choice questions. The highest possible score (with higher scores indicating more severe depression) is 63. The lowest possible score is 0.
Difference in scores for the Beck Anxiety Inventory between individuals with hearing loss and normal hearing controls. | 5 min
  The Beck Anxiety Inventory is a standard anxiety scale. It consists of a list of 21 anxiety symptoms and asks participants to indicate how much they have been bothered by each symptom by choosing from the following options: "Not At All", "Mildly", "Moderately", "Severely".

CONTACTS AND LOCATIONS:
Overall Officials: James E Saunders, MD, Principal Investigator — Department of Surgery, Otolaryngology section, Dartmouth Hitchcock Medical Center
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will be available to researchers involved in this study only.